CLINICAL TRIAL: NCT01418378
Title: A Double-blinded Randomised Controlled Trial Comparing the Performance of the Sigma® CR150 and Sigma® CR Knee Systems, When Used in Fixed Bearing Primary Cruciate Retaining Total Knee Arthroplasty for the Treatment of Osteoarthritis
Brief Title: Sigma CR150 Versus Sigma CR Knee RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT07/04
Record Dates: First submitted 2011-08-09; First posted 2011-08-17 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Osteoarthritis
Keywords: Sigma; cruciate; retaining; fixed; primary; total; knee; arthroplasty; cemented; osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sigma CR150 (Active Comparator): Sigma CR150 femoral component used in combination with the Highly Polished Cobalt Chrome fixed bearing tibial tray and the Curved (XLK) polyethylene bearing (cemented, no patellar resurfacing).
  Interventions: Device: Sigma CR150
- Sigma CR (Active Comparator): Sigma CR femoral component used in combination with the Highly Polished Cobalt Chrome fixed bearing tibial tray and the Curved (XLK) polyethylene bearing (cemented, no patellar resurfacing).
  Interventions: Device: Sigma CR

INTERVENTIONS:
Device: Sigma CR150 — Sigma CR150 femoral component used in combination with the Highly Polished Cobalt Chrome fixed bearing tibial tray and the Curved (XLK) polyethylene bearing (cemented, no patellar resurfacing).
  Other Names: PFC Sigma CR150
  Arms: Sigma CR150
Device: Sigma CR — Sigma CR femoral component used in combination with the Highly Polished Cobalt Chrome fixed bearing tibial tray and the Curved (XLK) polyethylene bearing (cemented, no patellar resurfacing).
  Other Names: PFC Sigma CR
  Arms: Sigma CR

SUMMARY:
This study will compare two very similar designs of knee replacement device. One device (Sigma CR150) is a slightly modified version of the original (Sigma CR) and has been modified to enhance/accommodate higher flexion. The original device has been in widespread clinical use with excellent results since 1996 and this study will determine whether the design modifications of the newer device add further value. The newer device has been in clinical use with good short-term(unpublished) outcomes since becoming commercially available in January 2009.

Achieving higher knee flexion may be required for cultural reasons or by the increasingly younger, more active patient population undergoing knee replacement today. In addition to promoting flexion, it is also possible that this design change may help the knee replacement to last longer than traditional implants in patients who achieve higher flexion. Therefore, the study will compare the two devices in terms of survivorship, flexion and other measures of the success of a total knee replacement (range of motion, knee-related quality of life, activity and generic quality of life) over the short-term.

A minimum of one hundred and forty subjects (minimum 70 per group) with osteoarthritis and aged 50-75 years will be included at UK/international hospitals.

Study duration is 2 years and patients will complete standard knee outcome scores plus radiological evaluation.

Subjects would receive one of the study devices regardless of their involvement in the study, and apart from (possible)additional visits, x-rays and/or questionnaires, treatment and follow-up care will be as per the care they would receive outside of the study.

ELIGIBILITY:
Inclusion Criteria:

i)Male or female subjects, aged between 50 and 75 years inclusive.

ii)Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.

iii) Subjects who, in the opinion of the Clinical Investigator, are able to understand this clinical investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

iv) Subjects defined by the Investigator as ASA Grade I or II.

v) Subjects with a primary diagnosis of osteoarthritis.

vi) Subjects who require a primary total knee arthroplasty.

vii) Subjects who can achieve active flexion of 90 degrees.

Exclusion Criteria:

i) Subjects who, in the opinion of the Clinical Investigator, have an existing condition that would compromise their participation and follow-up in this clinical investigation.

ii) Subjects who are known drug or alcohol abusers or with psychological disorders that could affect follow-up care or treatment outcomes.

iii) Subjects who have participated in a clinical investigation with an investigational product in the last month.

iv) Subjects who are currently involved in any injury litigation claims.

v) Subjects with an anatomical limb alignment of above 20 degrees varus or valgus.

vi) Subjects with a fixed flexion deformity of over 20 degrees.

vii) Subjects with recurvatum (definition: hyperextension ≥ 5 degrees).

viii) Subjects who cannot flex their hip to 90 degrees.

ix) Subjects with a BMI of 35 or above.

x) Subjects defined by the Investigator as ASA Grade III-V.

xi) Subjects who are identified pre-operatively as having bone defects which require augmentation.

xii) Subjects who have previously undergone total or unicondylar knee arthroplasty, high tibial osteotomy, ligament reconstruction, ORIF or with previous fracture in the knee joint.

xiii) Subjects with primary or secondary diagnosis of inflammatory or traumatic arthritis.

xiv) Subjects who have undergone contralateral total knee arthroplasty during the previous 6 months.

xv) Subjects who in the opinion of the Investigator require patellar resurfacing.

Intra-operative exclusion criteria:

i) Subjects who have uncontained bone defects or defects bigger than 8 mm3 and/or require augmentation.

ii) Subjects who are not suitable to receive both the study and comparator devices.

iii) Subjects who require patellar resurfacing

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2011-08-03 (Actual); Primary Completion 2016-02-17 (Actual); Study Completion 2016-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Chakrabarty, FRCS Orth., Principal Investigator — Calderdale and Huddersfield Foundation NHS Trust
Locations (4):
- Sunshine Hospitals, Secunderabad, Andhra Pradesh, India
- Singapore General Hospital, Singapore, Singapore
- United Kingdom (2):
  - Victoria Hospital, Kirkcaldy, Fife
  - Calderdale Royal Hospital, Halifax, West Yorkshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 191 subjects were recruited at sites in the UK, India and Singapore. Enrollment took place between 3 August 2011 and 21 January 2014
Pre-assignment Details: After written informed consent was obtained from subjects, eligibility was confirmed and subjects were allocated a subject identification number
Groups:
- Sigma CR 150: Subjects who received a Sigma CR 150 implant
- Sigma CR: Subjects who received a Sigma CR implant
Period: Overall Study
Arm/Group | Sigma CR 150 | Sigma CR
Started | 90 (A total of 191 subjects were enrolled into the study. 13/191 did not receive a study implant) | 88 (A total of 191 subjects were enrolled into the study. 13/191 did not receive a study implant)
Subjects Who Received Study Implant | 90 (the number of subjects implanted with study implant) | 88 (the number of subjects implanted with study implant)
Completed | 89 | 83
Not Completed | 1 | 5
Not completed — Death | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — ligament imbalance | 0 | 1
Not completed — developed chronic myopathy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sigma CR 150 | Sigma CR | Total
Number analyzed (Participants) | 90 | 88 | 178
Age, Continuous [Mean (Standard Deviation); unit: Years] — Subject age at time of consent
  Years | 63.2 (6.9) | 64.4 (6.2) | 63.8 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Subject gender
  Participants
    Female | 61 | 50 | 111
    Male | 29 | 38 | 67
Pre-operative flexion angle [Mean (Standard Deviation); unit: Degrees] — Pre-operative flexion angle was measured
  Degrees | 110.8 (21.4) | 110.4 (19.4) | 110.6 (20.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 27.1 (3.6) | 27.7 (3.9) | 27.4 (3.8)
Primary Diagnosis [Count of Participants; unit: Participants] — Subjects with primary diagnosis of osteoarthritis in the study knee
  Participants | 90 | 88 | 178

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Knees Who Survived at 2 Years Post-operative
Description: The Kaplan-Meier success rate at 24-months post-operatively was calculated with Kaplan-Meier time-to-event methodology, where the time variable for patients who were successful (no components revised for any reason) was censored at the time of last follow-up.
Time Frame: 2 Years
Population: Safety population
Measure: Number (95% Confidence Interval); unit: Percentage of Knees remaining
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 90 | 88
Percentage of Knees remaining | 100 [100 to 100] | 100 [100 to 100]

2. Secondary Outcome: Change From Baseline in Goniometer Measured Maximum Passive Flexion at 2 Years
Description: Comparative evaluation of the change from baseline values in 2 year goniometer-measured passive flexion. A goniometer is an instrument used to measure angles in degrees and captures the change in angle between the upper and lower leg
Time Frame: Pre-operative baseline to 2 years
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 73 | 63
degrees | -3.37 (12.97) | -0.67 (11.81)

3. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Pain Subscore - 1 Year
Description: Comparative evaluation of the change from baseline values at 1 years in Knee Injury and Osteoarthritis Outcome Pain Subscore
  The subscore ranges from 0 (no pain) to 36 (extreme pain). The subscore is then transformed into a 0 (extreme pain) to 100 (no pain) scale.
  100 - (score x 100) / 36 = transformed score
Time Frame: Pre-operative baseline to 1 year
Population: Subjects within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 75 | 61
Scores on a scale | 46.59 (16.68) | 48.54 (16.69)

4. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Pain Subscore - 2 Years
Description: Comparative evaluation of the change from baseline values at 2 years in Knee Injury and Osteoarthritis Outcome Pain Subscore
  The subscore ranges from 0 (no pain) to 36 (extreme pain). The subscore is then transformed into a 0 (extreme pain) to 100 (no pain) scale.
  100 - (score x 100) / 36 = transformed score
Time Frame: 2 years
Population: Study subjects at 2 years - Subjects within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 72 | 62
Scores on a scale | 51.50 (17.71) | 55.38 (15.40)

5. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Symptoms Subscore - 1 Years
Description: Comparative evaluation of the change from baseline values at 1 year in Knee Injury and Osteoarthritis Outcome Symptom Subscore
  The subscore ranges from 0 (no symptoms) to 36 (always have symptoms). The subscore is then transformed into a 0 (always have symptoms) to 100 (never have symptoms) scale.
  100 - (score x 100) / 36 = transformed score
Time Frame: 1 years
Population: Study subjects at 1 year - Subjects within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 75 | 61
Scores on a scale | 44.00 (20.95) | 39.99 (20.86)

6. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Symptom Subscore - 2 Years
Description: Comparative evaluation of the change from baseline values at 2 years in Knee Injury and Osteoarthritis Outcome Symptom Subscore
  The subscore ranges from 0 (never have symptoms) to 28 (always have symptoms). The subscore is then transformed into a 0 (always have symptoms) to 100 (never have symptoms) scale.
  100 - (score x 100) / 28 = transformed score
Time Frame: 2 years
Population: Study subjects at 2 year -Subjects within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 72 | 63
Scores on a scale | 38.59 (20.33) | 40.65 (18.17)

7. Secondary Outcome: Knee Injury and Osteoarthritis Outcome - Activities of Daily Living Subscore - 1 Years
Description: Comparative evaluation of the change from baseline values at 1 years in Knee Injury and Osteoarthritis Outcome Symptom Subscore
  The subscore ranges from 0 (no difficulty) to 68 (extreme difficulty). The subscore is then transformed into a 0 (extreme difficulty) to 100 (no difficulty) scale.
  100 - (score x 100) / 68 = transformed score
Time Frame: 1 year
Population: Study subjects at 1 year - Subjects within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 75 | 61
Scores on a scale | 44.00 (20.95) | 39.99 (20.86)

8. Secondary Outcome: Knee Injury and Osteoarthritis Outcome - Activities of Daily Living Subscore - 2 Years
Description: Comparative evaluation of the change from baseline values at 2 years in Knee Injury and Osteoarthritis Outcome Activities of Daily Living Subscore
  The subscore ranges from 0 (no difficulty) to 68 (extreme difficulty). The subscore is then transformed into a 0 (extreme difficulty) to 100 (no difficulty) scale.
  100 - (score x 100) / 68 = transformed score
Time Frame: 2 year
Population: Study subjects at 2 years - Subjects within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 72 | 63
Scores on a scale | 38.59 (20.33) | 40.65 (18.17)

9. Secondary Outcome: Knee Injury and Osteoarthritis Outcome - Sport and Recreation Subscore - 1 Years
Description: Comparative evaluation of the change from baseline values at 1 years in Knee Injury and Osteoarthritis Outcome Activities of Daily Living Subscore
  The subscore ranges from 0 (no difficulty) to 20 (extreme difficulty). The subscore is then transformed into a 0 (extreme difficulty) to 100 (no difficulty) scale.
  100 - (score x 100) / 20 = transformed score
Time Frame: 1 year
Population: Study subjects at 1 years - Subjects within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 73 | 60
Scores on a scale | 46.99 (32.82) | 46.42 (28.91)

10. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Sport and Recreation Subscore - 2 Years
Description: Comparative evaluation of the change from baseline values at 2 years in Knee Injury and Osteoarthritis Outcome Activities of Daily Living Subscore
  The subscore ranges from 0 (no difficulty) to 20 (extreme difficulty). The subscore is then transformed into a 0 (extreme difficulty) to 100 (no difficulty) scale.
  100 - (score x 100) / 20 = transformed score
Time Frame: 2 year
Population: Study subjects at 2 years - Subjects within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 70 | 63
Scores on a scale | 61.29 (35.60) | 60.40 (32.75)

11. Secondary Outcome: Knee Injury and Osteoarthritis Outcome - Quality of Life Subscore - 1 Years
Description: Comparative evaluation of the change from baseline values at 1 years in Knee Injury and Osteoarthritis Outcome Activities of Quality of life Subscore
  The subscore ranges from 0 (no difficulty) to 16 (extreme difficulty). The subscore is then transformed into a 0 (extreme difficulty) to 100 (no difficulty) scale.
  100 - (score x 100) / 16 = transformed score
Time Frame: 1 year
Population: Study subjects at 1 years - Subjects within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 75 | 61
Scores on a scale | 50.75 (24.83) | 49.59 (18.71)

12. Secondary Outcome: Knee Injury and Osteoarthritis Outcome - Quality of Life Subscore - 2 Years
Description: Comparative evaluation of the change from baseline values at 2 years in Knee Injury and Osteoarthritis Outcome Quality of Life Subscore
  The subscore ranges from 0 (no difficulty) to 16 (extreme difficulty). The subscore is then transformed into a 0 (extreme difficulty) to 100 (no difficulty) scale.
  100 - (score x 100) / 16 = transformed score
Time Frame: 2 years
Population: Study subjects at 2 years - Subjects within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 72 | 63
Scores on a scale | 60.33 (23.90) | 59.92 (21.23)

13. Secondary Outcome: Change From Baseline in Goniometer Measured Maximum Passive Flexion at 1 Year.
Description: Comparative evaluation of the change from baseline values in 1 year goniometer-measured passive Flexion. A goniometer is an instrument used to measure angles in degrees and captures the change in angle between the upper and lower leg. Passive flexion involves moving the leg through range of motion without active muscle contraction
Time Frame: 1 year
Population: Subjects at 1-year within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 74 | 62
degrees | -1.03 (12.65) | -0.23 (12.21)

14. Secondary Outcome: Change From Baseline in Goniometer Measured Maximum Passive Extension at 1 Year
Description: Comparative evaluation of the change from baseline values in 1 year goniometer-measured passive extension. A goniometer is an instrument used to measure angles in degrees and captures the change in angle between the upper and lower leg. Passive extension involves the leg being moved without active muscle contraction
Time Frame: 1 year
Population: Subjects at one year within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 74 | 62
degrees | -2.34 (4.84) | -3.15 (6.89)

15. Secondary Outcome: Change From Baseline in Goniometer Measured Maximum Passive Extension at 2 Years
Description: Comparative evaluation of the change from baseline values in 2 year goniometer-measured passive extension. A goniometer is an instrument used to measure angles in degrees and captures the change in angle between the upper and lower leg. Passive extension involves moving the leg without active muscle contraction
Time Frame: 2 year
Population: Subjects at 2 years within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 73 | 63
degrees | -2.63 (5.14) | -3.44 (7.78)

16. Secondary Outcome: Change From Baseline in Goniometer Measured Maximum Total Range of Motion at 1 Year
Description: Comparative evaluation of the change from baseline values in 1 year goniometer-measured total range of motion. A goniometer is an instrument used to measure angles in degrees and captures the change in angle between the upper and lower leg. Total range of motion is the full distance the lower leg travels in relation to the upper leg.
Time Frame: 1 year
Population: Subjects at 1 year within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 74 | 62
degrees | 1.31 (13.83) | 2.92 (14.59)

17. Secondary Outcome: Change From Baseline in Goniometer Measured Maximum Total Range of Motion at 2 Years.
Description: Comparative evaluation of the change from baseline values in 2 year goniometer-measured total range of motion. A goniometer is an instrument used to measure angles in degrees and captures the change in angle between the upper and lower leg. Total range of motion is the full distance the lower leg travels in relation to the upper leg.
Time Frame: 2 years
Population: Subjects at 2 years within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 73 | 63
degrees | -0.74 (14.42) | 2.78 (15.99)

18. Secondary Outcome: Number of Participants With Flexion Contracture at 1 Year
Description: Summary of flexion contracture at 1 year time point. Flexion contracture is a shortening of the muscles that prevents the leg from fully extending
Time Frame: 1 years
Population: Subjects at 1 year within per protocol population with complete, available data
Measure: Count of Participants; unit: Participants
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 75 | 62
Participants
  5-10 degrees | 7 | 5
  11-15 degrees | 1 | 0

19. Secondary Outcome: Number of Participants With Flexion Contracture at 2 Years
Description: Summary of flexion contracture at 2 year time point.Flexion contracture is a shortening of the muscles that prevents the leg from fully extending
Time Frame: 2 years
Population: Subjects at 2 years within per protocol population with complete, available data
Measure: Count of Participants; unit: Participants
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 77 | 65
Participants
  5-10 degrees | 4 | 2
  11-15 degrees | 0 | 0

20. Secondary Outcome: Total Knee Society Score at 1 Year
Description: Total Knee Society Knee Score change from baseline at 1 year
  The Total Knee Society Score is comprised of two scores: the Knee Score and the Function Score. Both have a 0-100 range. Sub-scales are combined to compute a total score of 100
  The Total Knee Society Score is made up of pain, range of motion, alignment and stability subscores. An Excellent score is 80-100, a good score is 70-79, a fair score is 60-69 and a poor score is anything below 60.
Time Frame: 1 year
Population: Subjects at 1 year within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 74 | 62
Scores on a scale | 45.07 (17.99) | 52.50 (14.76)

21. Secondary Outcome: Total Knee Society Knee Score at 2 Years
Description: Total Knee Society Knee Score change from baseline at 2 years
  The Total Knee Society Score is comprised of two scores: the Knee Score and the Function Score. Both have a 0-100 range. Sub-scales are combined to compute a total score of 100
  The Total Knee Society Score is made up of pain, range of motion, alignment and stability subscores. An Excellent score is 80-100, a good score is 70-79, a fair score is 60-69 and a poor score is anything below 60.
Time Frame: 2 years
Population: Subjects at 2 years within per protocol population with complete, available data
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 73 | 63
Scores on a scale | 46.44 (17.74) | 54.51 (15.71)

22. Secondary Outcome: Anatomic Alignment Angle
Description: Anatomic angle measured at 1 year time point.
  If one draws a line from the center of the hip joint to the center of the ankle joint this is considered to be the mechanical axis of the femur.
  A line drawn through the center of the femoral shaft is the anatomic axis.
  The angle created at the intersection of these lines is referred to as the anatomic alignment angle.
  A normal angle is approximately 7-9 degrees "valgus" or slightly "knock-kneed". "Varus" angles are less common and are also referred to as "bow-legged".
Time Frame: 1 year time point
Population: Subjects at 1 year within safety population with complete, available data
Measure: Count of Participants; unit: Participants
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 67 | 67
Participants
  Varus | 1 | 0
  valgus | 66 | 67

23. Secondary Outcome: Anatomic Alignment Angle
Description: Anatomic angle measured at 2 year time point.
  If one draws a line from the center of the hip joint to the center of the ankle joint this is considered to be the mechanical axis of the femur.
  A line drawn through the center of the femoral shaft is the anatomic axis.
  The angle created at the intersection of these lines is referred to as the anatomic alignment angle.
  A normal angle is approximately 7-9 degrees "valgus" or slightly "knock-kneed". "Varus" angles are less common and are also referred to as "bow-legged".
Time Frame: 2 year time point
Population: Subjects at 2 years within safety population with complete, available data
Measure: Count of Participants; unit: Participants
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 69 | 65
Participants
  Varus | 3 | 0
  Valgus | 66 | 65

24. Secondary Outcome: Alignment - Femoral Component to Anatomic Angle.
Description: Femoral component angle measured at 1 year time point. This angle is measured between a line drawn from the center of the femoral head and a line across the bottom of the femoral implant (condyles).
Time Frame: 1 year time point
Population: Subjects at 1 year within safety population with complete, available data
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 82 | 79
Degrees | 94.37 (1.95) | 94.21 (2.64)

25. Secondary Outcome: Alignment - Femoral Component to Anatomic Angle
Description: Femoral component angle measured at 2 year time point. This angle is measured between a line drawn from the center of the femoral head and a line across the bottom of the femoral implant (condyles).
Time Frame: 2 year time point
Population: Subjects at 2 year within safety population with complete, available data
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 80 | 77
Degrees | 93.94 (2.11) | 94.48 (2.2)

26. Secondary Outcome: Alignment - Tibial Component to Anatomic Angle
Description: Tibial component angle measured at 1 year time point. This angle is measured between a line drawn from the center of the femoral head tibial implant.
Time Frame: 1 year time point
Population: Subjects at 1 year within safety population with complete, available data
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 82 | 80
Degrees | 89.96 (1.39) | 90.06 (1.83)

27. Secondary Outcome: Alignment - Tibial Component to Anatomic Angle
Description: Tibial component angle measured at 2 year time point. This angle is measured between a line drawn from the center of the femoral head tibial implant.
Time Frame: 2 year time point
Population: Subjects at 2 year within safety population with complete, available data
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 80 | 77
Degrees | 89.69 (1.60) | 90.19 (1.98)

28. Secondary Outcome: Alignment - Femoral Component Flexion
Description: Femoral Component Flexion measured at 1 year time point. This measures the angle between a line drawn though the center of the side of the femur and a line drawn across the top of the flat inner surface of the femoral component.
Time Frame: 1 year time point
Population: Subjects at 1 year within safety population with complete, available data
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 82 | 80
Degrees | 89.74 (2.44) | 90.10 (2.12)

29. Secondary Outcome: Alignment - Femoral Component Flexion
Description: Alignment - Femoral Component Flexion measured at 2 year time point. This measures the angle between a line drawn though the center of the side of the femur and a line drawn across the top of the flat inner surface of the femoral component.
Time Frame: 2 year time point
Population: Subjects at 2 years within safety population with complete, available data
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 80 | 77
Degrees | 89.93 (2.35) | 89.80 (2.99)

30. Secondary Outcome: Alignment - Tibial Posterior Slope
Description: Tibial Posterior Slope measured at 1 year time point. This angle is measured between a line through the center of the side of the tibia and the top flat surface of the tibial implant
Time Frame: 1 year time point
Population: Subjects at 1 year within safety population with complete, available data
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 82 | 80
Degrees | 85.95 (2.25) | 85.47 (2.62)

31. Secondary Outcome: Alignment - Tibial Posterior Slope
Description: Alignment - Tibial Posterior Slope measured at 2 year time point. This angle is measured between a line through the center of the side of the tibia and the top flat surface of the tibial implant
Time Frame: 2 year time point
Population: Subjects at 2 years within safety population with complete, available data
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 80 | 76
Degrees | 85.99 (2.29) | 85.15 (3.24)

32. Secondary Outcome: Number of Subjects With Radiolucencies - Femoral Component
Description: The bone-implant interface at the femoral components were examined radiographically and radiolucencies were measured in millimeters.
  Radiolucent lines (RLLs) greater than 2mm are considered to be clinically significant.
Time Frame: 6 to 12 week and 24 month intervals
Population: Subjects within safety population with complete, available data
Measure: Count of Participants; unit: Participants
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 90 | 88
Participants
  6 Weeks to 12 Weeks | 0 | 2
  24 months | 2 | 1

33. Secondary Outcome: Number of Subjects With Radiolucencies - Tibial Component
Description: The bone-implant interface at the tibial components were examined radiographically and radiolucencies were measured in millimeters.
  Radiolucent lines (RLLs) greater than 2mm are considered to be clinically significant.
  Radiolucent lines greater than 2mm are considered to be clinically significant.
Time Frame: 6 weeks to 24 months
Population: Subjects within safety population with complete, available data
Measure: Count of Participants; unit: Participants
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 90 | 88
Participants
  6 Weeks to 12 Weeks | 0 | 1
  12 months | 0 | 1

34. Secondary Outcome: Radiographic Evaluation of Maximum Flexion
Description: Maximum knee flexion measured radiographically at 1 year time point
Time Frame: 1 year time point
Population: Subjects at 1 year within safety population with complete, available data
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Sigma CR 150 | Sigma CR
Number analyzed (Participants) | 74 | 70
Degrees | 108.51 (18.90) | 107.11 (17.41)

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events were evaluated during clinic visits at protocol-defined post-operative intervals
Groups:
- CR 150: Subjects who received a Sigma CR150 implant
- C-RET: Subjects who received a Sigma CR implant
Arm/Group | CR 150 | C-RET
Serious Adverse Events (participants affected / at risk) | 9/90 | 8/88
Other Adverse Events (participants affected / at risk) | 14/90 | 14/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CR 150 (N=90) | C-RET (N=88)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CR 150 (N=90) | C-RET (N=88)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 (14) | 14 (14)

LIMITATIONS AND CAVEATS:
Many subjects had last visit before 2yrs from date of surgery-KM survivorship estimate calculated at 1.8 years when 40 knees left in study. Subject data not available for every outcome- numbers analyzed vary between outcomes and Participant Flow.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less